CLINICAL TRIAL: NCT01473030
Title: Long-term Effects of Dutasteride on Architectural and Nuclear Morphometric Features of Benign Prostate Tissue
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Peter Gann, Professor and Director, Division of Pathology Research, University of Illinois at Chicago
Other Study IDs: 2011-0646
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Benign Prostate Tissue
Keywords: Benign prostate; serum DHT; Dutasteride; PSA; Avodart

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Biopsy tissue (Year 2 and Year 4) already collected in REDUCE trial
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dutasteride: No PCa at Year 2 or Year 4
- Placebo: No PCa at Year 2 or Year 4

SUMMARY:
The overall goal of this project is to quantify the long-term effects of dutasteride on the architectural and nuclear features of benign prostate tissue, using state-of-the art digital image analysis techniques. The ultimate result will be a multivariable morphological "signature" that could provide a useful indicator of an individual's degree of drug response.

ELIGIBILITY:
Inclusion Criteria:

* completed REDUCE trial (Year 4 exit biopsy with blocks and HE slides available; i.e., U.S. participants only)
* compliant with assigned treatment based on either: (dutasteride group) at least 3 post-baseline serum DHT levels ≥ 50% lower than baseline, or (placebo group) at least 3 post-baseline serum DHT levels with none showing ≥ 50% decrease from baseline
* subgroup: Year 2 biopsy blocks and HE slides available for Aim 4a

Exclusion Criteria:

* N/A

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cross-sectional comparison of biomarkers in prostate biopsy tissue (Year 2 and Year 4) already collected in REDUCE trial
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Architectural Features | Year 4
  To characterize and quantify the effects of dutasteride on histological (architectural) features of benign prostate tissue via comparison of a random sample of Year 4 biopsy specimens from the dutasteride and placebo groups.
Morphometric features | Year 4
  To quantify the long-term (Year 4) effects of dutasteride on nuclear morphometric features (i.e., size, shape and texture) in benign prostatic epithelial cells.
  To develop and validate a multivariable morphological score based on summarization of differences between drug- and placebo-treated tissues.
Independent changes in architecture and morphometry | Year 4
  To determine the degree to which drug-related changes at Year 4 in architectural and nuclear features are independent of (i.e., not explained by) changes in serum DHT, gland volume and PSA.

SECONDARY OUTCOMES:
Changes in cytomorphology | Year 2 & Year 4
  To determine, by comparing Year 2 to Year 4 samples within individuals, whether drug-related cytomorphological changes are constant, declining or progressing.

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Gann, MD, ScD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States